CLINICAL TRIAL: NCT03584464
Title: A Post-approval Study of the Medtronic Resolute Onyx™ Zotarolimus-Eluting Coronary Stent System
Brief Title: RESOLUTE ONYX Post-Approval Study (Bifurcation Cohort)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Ver 4.0 16Feb2018
Record Dates: First submitted 2018-05-14; First posted 2018-07-12 (Actual); Results first posted 2022-01-12 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Bifurcation Cohort (Other): Subjects receiving stents 2.0 mm - 5.0 mm in diameter will be included in the Bifurcation Cohort.
  Interventions: Device: Resolute Onyx™ Zotarolimus-Eluting Coronary Stent System

INTERVENTIONS:
Device: Resolute Onyx™ Zotarolimus-Eluting Coronary Stent System — Medtronic Resolute Onyx™ Zotarolimus-Eluting Coronary Stent System, sizes 2.0 mm - 5.0 mm

SUMMARY:
To observe the continued performance of the Medtronic Resolute Onyx™ Zotarolimus-Eluting Coronary Stent System in a real-world more-comer population.

To collect data on the safety and efficacy of the Medtronic Resolute Onyx™ Zotarolimus-Eluting Coronary Stent System in bifurcated lesions.

ELIGIBILITY:
Key Inclusion Criteria

* Symptomatic coronary artery disease including subjects with chronic stable angina, silent ischemia, and acute coronary syndromes including non-ST elevation and ST-elevation myocardial infarction
* Subject is an acceptable candidate for treatment with a drug eluting stent in accordance with the applicable guidelines on percutaneous coronary interventions, manufacturer's Instructions for Use, and the Declaration of Helsinki
* Subject requires treatment of a single de novo bifurcated lesion amenable to treatment with Resolute Onyx using the provisional stenting technique

Exclusion Criteria:

* Unprotected left main disease
* Subjects with planned PCI of three vessel disease
* Planned two stent technique (main branch and side branch) of a bifurcation
* Subjects with more than one bifurcation lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2022-09-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (21):
  - Huntsville Hospital, Huntsville, Alabama
  - Scripps Green Hospital, La Jolla, California
  - Riverside Community Hospital, Riverside, California
  - Hartford Hospital, Hartford, Connecticut
  - Morton Plant Hospital, Clearwater, Florida
  - North Florida Regional Medical Center, Gainesville, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - WellStar Kennestone Hospital, Marietta, Georgia
  - University of Michigan Health System, Ann Arbor, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Abbott Northwestern, Minneapolis, Minnesota
  - Nebraska Medical Center, Omaha, Nebraska
  - Desert Springs Hospital, Las Vegas, Nevada
  - St. Josephs Hospital Health Center, East Syracuse, New York
  - North Shore University Hospital, Manhasset, New York
  - NYU Langone Medical Center, New York, New York
  - New York-Presbyterian Hospital/ Columbia University Medical Center, New York, New York
  - Baptist Memorial Hospital-Memphis, Germantown, Tennessee
  - Houston Methodist Hospital, Houston, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Saint Vincent Hospital, Green Bay, Wisconsin
- Belgium (2):
  - CHU Charleroi, Charleroi
  - Ziekenhuis Oost Limburg, Genk
- CHU Toulouse - Hôpital Rangueil, Toulouse, France
- Stredoslovensky Ustav Srdcovych a Cievnych Chorob a.s, Banská Bystrica, Slovakia

RESULTS

PARTICIPANT FLOW:
Groups:
- Bifurcation Cohort: Subjects receiving stents 2.0 mm - 5.0 mm in diameter will be included in the Bifurcation Cohort.
  Resolute Onyx™ Zotarolimus-Eluting Coronary Stent System: Medtronic Resolute Onyx™ Zotarolimus-Eluting Coronary Stent System, sizes 2.0 mm - 4.0 mm
Period: Overall Study
Arm/Group | Bifurcation Cohort
Started | 205
Completed | 204 (Number of subjects that competed 1 year follow up or had a CEC event)
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Bifurcation Cohort: Subjects receiving stents 2.0 mm - 5.0 mm in diameter will be included in the Bifurcation Cohort.
  Resolute Onyx™ Zotarolimus-Eluting Coronary Stent System: Medtronic Resolute Onyx™ Zotarolimus-Eluting Coronary Stent System, sizes 2.0 mm - 5.0 mm in diameter for the treatment of a bifurcation lesion with provisional stenting.
Arm/Group | Bifurcation Cohort
Number analyzed (Participants) | 205
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 87
  >=65 years | 118
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 161
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Subjects did not provide this information
  Participants
    number analyzed (Participants) | 194
    Hispanic or Latino | 12
    Not Hispanic or Latino | 182
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Subjects did not provide this information
  Participants
    number analyzed (Participants) | 193
    American Indian or Alaska Native | 0
    Asian | 8
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 11
    White | 159
    More than one race | 15
    Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 167
  Europe | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: Target Vessel Failure (TVF) defined as cardiac death, target vessel myocardial infarction, or clinically-driven target vessel revascularization by percutaneous or surgical methods.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Bifurcation Cohort
Number analyzed (Participants) | 204
Participants | 14

2. Secondary Outcome: Number of Participants With Cardiac Death
Description: Cardiac Death defined as any death due to immediate cardiac cause, unwitnessed death and death of unknown cause.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bifurcation Cohort
Number analyzed (Participants) | 204
Participants | 3

3. Secondary Outcome: Number of Participants With Target Vessel Myocardial Infarction (TVMI - 3rd UDMI)
Description: Target Vessel Myocardial Infarction (TVMI) defined as myocardial infarction with the target vessel. (3rd UDMI)
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bifurcation Cohort
Number analyzed (Participants) | 204
Participants | 6

4. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: Target Lesion Revascularization (TLR) defined as repeat PCI (Percutaneous Coronary Intervention), CABG (Coronary Artery Bypass Surgery) to the target lesion, or clinically driven target lesion revascularization.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bifurcation Cohort
Number analyzed (Participants) | 204
Participants | 7

5. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: Target Vessel Revascularization (TVR) defined as revascularization of the target vessel.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bifurcation Cohort
Number analyzed (Participants) | 204
Participants | 8

6. Secondary Outcome: Number of Participants With Cardiac Death and TVMI
Description: Cardiac Death and TVMI defined as composite of cardiac death and target vessel myocardial infarction.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bifurcation Cohort
Number analyzed (Participants) | 204
Participants | 9

7. Secondary Outcome: Number of Participants With Major Adverse Cardiac Event (MACE)
Description: Major Adverse Cardiac Event (MACE) defined as death, myocardial infarction (Q wave and non-Q wave), emergent coronary bypass surgery, or clinically driven repeat target lesion revascularization by percutaneous or surgical methods.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bifurcation Cohort
Number analyzed (Participants) | 204
Participants | 17

8. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: Target Lesion Failure (TLF) defined as cardiac death, target vessel myocardial infarction (Q wave and non-Q wave), or clinically driven target lesion revascularization (TLR) by percutaneous or surgical methods.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bifurcation Cohort
Number analyzed (Participants) | 204
Participants | 13

9. Secondary Outcome: Number of Participants With Stent Thrombosis (ARC) Definite/Probable
Description: Stent Thrombosis Definite/Probable defined per Academic Research Consortium (ARC).
  Definite: a. Angiographic confirmation of TIMI flow grade 0-3 and at least one of the following criteria within a 48 hour: 1.New onset s ischemic symptoms at rest (typical chest pain with duration >20 minutes); 2.New ischemic ECG changes suggestive of acute ischemia; 3.Typical rise and fall in cardiac biomarkers. or b. Pathologic confirmation of stent thrombosis: Evidence of recent thrombus within the stent determined at autopsy or via examination of tissue retrieved following thrombectomy.
  Probable: Any unexplained death within the first 30 days.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bifurcation Cohort
Number analyzed (Participants) | 204
Participants | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Bifurcation Cohort
All-Cause Mortality (participants affected / at risk) | 6/205
Serious Adverse Events (participants affected / at risk) | 48/205
Other Adverse Events (participants affected / at risk) | 39/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bifurcation Cohort (N=205)
Normocytic Anaemia (Blood and lymphatic system disorders) | 1 (1)
Acute Left Ventricular Failure (Cardiac disorders) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 4 (4)
Angina Pectoris (Cardiac disorders) | 4 (4)
Angina Unstable (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 2 (2)
Atrioventricular Block Second Degree (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 2 (2)
Cardiac Failure Congestive (Cardiac disorders) | 2 (3)
Coronary Artery Disease (Cardiac disorders) | 4 (4)
Coronary Artery Dissection (Cardiac disorders) | 1 (1)
Sinus Arrest (Cardiac disorders) | 1 (1)
Diverticulum Intestinal (Gastrointestinal disorders) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (2)
Melaena (Gastrointestinal disorders) | 1 (2)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Death (General disorders) | 1 (1) — Site reported an unknown cause of death, therefore there is no known event that led to death. The event has been reviewed by our Safety Specialist and was adjudicated.
Non-Cardiac Chest Pain (General disorders) | 1 (1)
Vascular Stent Stenosis (General disorders) | 1 (1)
Vessel Puncture Site Haematoma (General disorders) | 1 (1)
Drug Hypersensitivity (Immune system disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Localised Infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 2 (2)
Septic Shock (Infections and infestations) | 1 (1)
Cardiac Procedure Complication (Injury, poisoning and procedural complications) | 1 (1)
Postoperative Respiratory Failure (Injury, poisoning and procedural complications) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1)
Myocardial Necrosis Marker Increased (Investigations) | 3 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Unresponsive To Stimuli (Nervous system disorders) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Carotid Endarterectomy (Surgical and medical procedures) | 1 (1)
Coronary Artery Bypass (Surgical and medical procedures) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bifurcation Cohort (N=205)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Blood Loss Anaemia (Blood and lymphatic system disorders) | 1 (1)
Angina Pectoris (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Bundle Branch Block Left (Cardiac disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 3 (3)
Coronary Artery Dissection (Cardiac disorders) | 2 (2)
Coronary Artery Occlusion (Cardiac disorders) | 1 (1)
Left Ventricular Dysfunction (Cardiac disorders) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 1 (1)
Gingival Bleeding (Gastrointestinal disorders) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1)
Chest Discomfort (General disorders) | 1 (1)
Chest Pain (General disorders) | 2 (2)
Injection Site Haemorrhage (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Vascular Stent Stenosis (General disorders) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Cardiac Procedure Complication (Injury, poisoning and procedural complications) | 1 (1)
Face Injury (Injury, poisoning and procedural complications) | 1 (1)
Patella Fracture (Injury, poisoning and procedural complications) | 1 (1)
Periprocedural Myocardial Infarction (Injury, poisoning and procedural complications) | 1 (1)
Plaque Shift (Injury, poisoning and procedural complications) | 1 (1)
Vascular Access Complication (Injury, poisoning and procedural complications) | 1 (1)
Vascular Access Site Swelling (Injury, poisoning and procedural complications) | 1 (1)
Inflammatory Marker Increased (Investigations) | 1 (1)
Myocardial Necrosis Marker Increased (Investigations) | 7 (7)
Troponin I Increased (Investigations) | 1 (1)
Troponin Increased (Investigations) | 3 (3)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Labile Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/64/NCT03584464/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-10): https://cdn.clinicaltrials.gov/large-docs/64/NCT03584464/SAP_001.pdf